CLINICAL TRIAL: NCT02932124
Title: Application of Mechanical Cardiopulmonary Resuscitation Devices and Their Value in Out-of-hospital Cardiac Arrest: A Retrospective Analysis of the German Resuscitation Registry
Status: Completed | Type: Observational
Sponsor: German Resuscitation Registry (Other)
Responsible Party: Principal Investigator, Jan-Thorsten Graesner, MD, PD Dr., German Resuscitation Registry
Other Study IDs: GRR-CC07-14
Record Dates: First submitted 2016-10-06; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Out-of-hospital Cardiac Arrest
Keywords: German Resuscitation Registry; out-of-hospital cardiac arrest; cardiopulmonary resuscitation; mechanical chest compression devices
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: manual chest compressions
- 2: mechanical chest compression
  Interventions: Device: mechanical chest compression device

INTERVENTIONS:
Device: mechanical chest compression device
  Groups: 2

SUMMARY:
The aim of this study was to analyse a large CPR database, the German Resuscitation Registry, to evaluate potential benefits of mechanical CPR devices over manual CPR in adult cardiac arrest victims. The primary endpoint considered is ROSC.

DETAILED DESCRIPTION:
In a retrospective analysis of the German Resuscitation Registry between 2007-2014, investigators examined the outcome after using mechanical CPR on return of spontaneous circulation (ROSC) in adults with out-of-hospital cardiac arrest (OHCA). Investigators compared mechanical CPR (Intervention group) to manual CPR (control group). According to preclinical risk factors, investigators calculated the predicted ROSC-after-cardiac-arrest (RACA) score for each group, and compared it to the rate of ROSC observed. Using multivariate analysis, investigators adjusted the influence of the devices' application on ROSC for epidemiological factors and therapeutic measures.

ELIGIBILITY:
Inclusion Criteria:

* out of hospital cardiac arrest
* during time prod from January 2007 until December 2014
* CPR attempted

Exclusion Criteria:

* Investigators excluded cases in which CPR was continued for less than five minutes, or duration of CPR was missing, as the outcome in this early period is not affected by the CPR mode.
* Children aged less than 18 years and patients of unknown age were also excluded as the devices are not approved for resuscitation on children.
* An active compression-decompression (ACD) is a hand-held suction device, to compress and actively decompress the chest after each compression.
* Investigators also excluded cases where ACD CPR was used, because it constitutes a different technology.
* Cases due to trauma were excluded as application of mechanical CPR devices may be limited due in traumatic events.
* Cases where data on ROSC and/or CPR mode was missing were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient suffering OHCA and be resuscitated by EMS where the data were delivered to the German Resuscitation Registry
Sampling Method: Non-Probability Sample
Enrollment: 19609 (Actual)
Dates: Start 2007-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
return of spontaneous circulation | sustained ROSC at any time latest after 24 hours
  sustained return of spontaneous circulation at any time during CPR

CONTACTS AND LOCATIONS:
Overall Officials: Jan Wnent, MD, Principal Investigator — German Resuscitation Registry

IPD SHARING:
Plan to Share IPD: No